CLINICAL TRIAL: NCT04170647
Title: Reperfusion Rates of Intravenous Tissue-type Plasminogen Activator on Acute Ischemic Stroke Patients With Large Vessel Occlusions and Predictor Factors of Recanalization
Brief Title: Efficacy of Intravenous Tissue-type Plasminogen Activator on Acute Ischemic Stroke Patients With Large Vessel Occlusions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Tinh Quang DANG, MD, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: UMP11192019
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Stroke, Ischemic; Stroke, Acute
Keywords: reperfusion; IVT
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Plasminogen Activators

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Plasminogen Activators — standard dosage of 0.9 mg/kg or reduced dosage of 0.6 mg/kg, divided into a 15% bolus and an 85% venous infusion

SUMMARY:
This is an observational prospective study about the reperfusion rate of intravenous thrombolysis on ischemic stroke patients with large vessel occlusions and predictor factors of successful recanalization.

DETAILED DESCRIPTION:
Stroke is one the most common cause of mortality and disabilities in the world, with the highest incidence in East Asia. Current American Stroke Association (ASA) and European Stroke Organisation (ESO) guidelines recommend bridging therapy with IVT for all eligible patients before indicating endovascular thrombectomy (EVT) for those with large vessel occlusions (LVO). Nevertheless, the decision to use IVT on stroke patients with LVO is still debatable, with many arguments against and supporting combined therapy or direct mechanical thrombectomy. At present, guideline in our hospital advocates the use of IVT in all patients who meet eligibility criteria and present within the 4,5 hour window for anterior circulation stroke and within 24 hour window for posterior circulation stroke. Due to the overcrowded nature of our center as a high-end specialization establishment in Vietnam, it is noted that our door-to-groin time is sub-optimal. This fact inadvertently prolongs the time of action of intravenous tissue-type plasminogen activator before the re-assessment of occlusion site on interventional radiography. Therefore, it is possible for us to better estimate the reperfusion effectiveness of IVT as well as analyse other factors that might have an influence on this rate. The goal of our study is to determine the recanalization rate of IVT and related predictor factors in AIS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older with consent form signed.
2. Patients hospitalized in 115 People's Hospital for acute ischemic stroke.
3. Patients receiving full dose of IVT, with a confirmed LVO (including MCA M1, MCA M2, ICA, BA and VA) on angiography and repeat vascular imaging within 24 hours of hospitalization.

Exclusion Criteria:

1. Patients with evidence of chronic occlusion of large vessels.
2. Patients without source angiography data to assess the characteristics of thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients presented at our hospital with LVO confirmed who received both intravenous tissue-type plasminogen activator and subsequent repeat angiography will be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
reperfusion rate | within 24 hours of hospitalization
  the reperfusion rate of intravenous thrombolysis in acute ischemic stroke with large vessel occlusion first confirmed by angiography and assessed later by a vascular imaging modality.

SECONDARY OUTCOMES:
symptomatic intracerebral hemorrhage | 48 hours after initiation of IVT
  incidence of symptomatic intracerebral hemorrhage 48 hours after initiation of IVT

CONTACTS AND LOCATIONS:
Locations (1):
- 115 People's Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided